CLINICAL TRIAL: NCT03198936
Title: Effect of Brain Pill™ on Working Memory Capacity and Mood Behaviour in Healthy Adults With Subjective Memory Complains and Mild Mood Disturbances.
Brief Title: To Access the Effect of Brain Pill™ on Working Memory Capacity and Mood Behaviour.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Leading Edge Marketing LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: LM/161103/BP/MCI
Record Dates: First submitted 2017-04-06; First posted 2017-06-26 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Memory Dysfunction; Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognizin® SynapsaTM (Experimental): Dose - 2 capsules twice a day with meals
  Interventions: Dietary Supplement: Cognizin® SynapsaTM
- Placebo (Placebo Comparator): Matching placebo capsules with microcrystalline cellulose with added colours Dose - 2 capsules twice a day with meals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cognizin® SynapsaTM — 2 capsules to be taken twice a day with meals with a glassful of water
  Arms: Cognizin® SynapsaTM
Dietary Supplement: Placebo — 2 capsules to be taken twice a day with meals with glassful of water
  Arms: Placebo

SUMMARY:
Brain Pill™ is a mental health enhancing and successfully marketed dietary supplement.

DETAILED DESCRIPTION:
Brain Pill™ is a mental health enhancing and successfully marketed dietary supplement with a balanced composition of scientifically proven nutrients for accelerating and restoring brain function and thereby enhancing the cognitive performance and creating positive impact on behavioral outcomes.Hence the aim of the study is assessment of the effects of Brain Pill supplementation on memory performance in healthy adults with subjective memory complaints.

It is a double-blind, randomized, placebo-controlled , single centered study to access the efficacy of Brain Pill on working memory capacity and mild mood disturbances.

Effect of Brain Pill on working memory capacity will be accessed by improvement in mean response time and accuracy measured by working memory battery from baseline to end of the study. Effect of Brain Pill is also accessed on Neurophysiological improvement in working memory as measured by electroencephelogram (EEG) from baseline to end of the study. Also improvement in attention and concentration will be accessed from baseline to end of the study by Picture recognition test.

Effect of Brain Pill on mood disturbances will be accessed by Brunel Universal Mood State.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Mini-Mental State Examination (MMSE) score > 23 indicating a healthy cognitive state.
* Subjects with Adult Memory Questionnaire (AMQ) score of 40-70% indicating subjective memory lapse.
* Subjects with T score on 8-item Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form: 50.0-59.9 (mild) as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM -5) criteria.
* Males and Females of Age 18 - 60 years will be selected for the study.
* Subject who is willing to maintain his or her habitual diet and usual physical activity patterns throughout the study.
* Subject who has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
* Subject should be willing to refrain from consuming alcohol 24 h prior to the test days.
* Subject should be willing to refrain from consuming caffeine and caffeine-containing products 12 h prior to test days.
* Subject should be willing to refrain from vigorous physical activity 12 h prior to test days.
* Subject should be a non-smoker.
* Subject who understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subjects with MMSE score ≤ 23 indicative of clinical dementia.
* Subjects with AMQ score <40 and >70 %.
* T score on 8-item PROMIS Depression Short Form <50 (normal) and ≥60 (moderate and severe).
* Confirmed diagnosis of dementia/ Alzheimer's disease.
* Current evidence of hearing impairment or other information processing impairment.
* Subjects who are using amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, 3,4-methylenedioxymethamphetamine, opiates or tricyclic antidepressants, as disclosed at the screening visit.
* Subjects with uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the average blood pressure measured at the screening.
* Subjects with a history or presence of clinically important cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorders that, in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
* Subject with a history, in the judgment of the Investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study or which could significantly influence cognitive abilities.
* Use of any sleep aid medication.
* Pregnant female subjects or planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Excessive habitual caffeine consumption (>300 mg caffeine/d or ≥3 cups of caffeinated coffee/d), following screening and throughout the study period.
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Use of antibiotics or signs of active systemic infection. Treatment visits will be rescheduled to allow the subject to wash off of the antibiotic for at least five days prior to any test visit.
* Subject who has had exposure to any non-registered drug product within 30 days prior to the screening visit.
* Subjects who are using any dietary supplements and or containing any of the ingredients of the investigational product.
* Recent history of (within 12 months of screening visit 1) or strong potential for alcohol or substance abuse.(Alcohol abuse is defined as >14 drinks per week.)
* Subject who has a known allergy or sensitivity to the study product or any ingredients of the study product or meals provided.
* The subject is unable to perform the tests on the computer for participation in this type of study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Working Memory Capacity | 84 days
  To evaluate effect of Brain Pill™ on working memory capacity as improvement in mean response time and accuracy and measured by working memory battery.

SECONDARY OUTCOMES:
Attention and Concentration | 84 days
  To evaluate effect of Brain Pill™ on attention and concentration as measured by Picture recognition test (PRT).
Improvement in Mood Disturbances | 84 days
  To evaluate effect of Brain Pill™ on mood disturbances as measured by Brunel Universal Mood States (BRUMS).

CONTACTS AND LOCATIONS:
Overall Officials: Divya Patel, BSc, Study Chair — Affiliated
Locations (1):
- Vedic Lifesciences Pvt.Ltd, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No